CLINICAL TRIAL: NCT05632952
Title: Laparoscopic Ventral Hernia Repair in Obese Patients: Safe and Effective Use of a Hybrid (PTFE / Biosynthetic) Mesh. Results of a Multicentric Prospective Trial.
Brief Title: ProSpectic Italian Laparoscopic Hybrid mEsh hErnia Repair in Obese patientS Trials
Acronym: PSICHE-EROS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, PhD, Md, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 419N.Reg 26-2022oss
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Uncomplicated Ventral Incisional Hernia; Obesity
Keywords: IPOM Plus,; incisional Hernia; Ventral Hernia; Obesity
MeSH Terms: conditions — Obesity; Incisional Hernia; Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- A: 120 patients affected by Incisional Hernia with size between 3 to 10 cm, undergoing Intraperitoneal Onlay Mesh with the closure of defect
  Interventions: Device: Intraperitoneal Onlay Mesh positioning Plus

INTERVENTIONS:
Device: Intraperitoneal Onlay Mesh positioning Plus — Intraperitoneal Onlay Mesh (IPOM) Plus with closure of the hernia defect will be performed according to the common recommendations.
  The closure of the wall defect will be decided according to the surgeon evaluations: hernia size and choice of technique will be recorded in the database. The mesh will have an overlap of at least 5 cm on all sides of the defect. Dimension of the mesh will be sized to overlap the hernia orifice by at least five centimetres and placed in the intraperitoneal position. Using non-articulating laparoscopic fixation devices, 5.1-mm non-absorbable or absorbable tacks will be then positioned around the circumference of the prosthesis in a 3-row manner or 2-row manner based on the intraoperative findings, the patient's specific situation and the operating surgeon's decision.
  Other Names: IPOM plus

SUMMARY:
The aim of this study is to evaluate safety and effectiveness of a hybrid mesh (GORE® SYNECOR Intraperitoneal Biomaterial) in patients with a BMI of 30 kg/m2 or more undergoing laparoscopic ventral hernia repair (LVHR) with intraperitoneal position of the mesh.

DETAILED DESCRIPTION:
A prospective Italian multicenter observational trial will be conducted in 8 different Italian centers to compare the effectiveness and feasibility of treatment of Incisional Hernia with GORE® SYNECOR Intraperitoneal Biomaterial mesh in patients with BMI >30 kg/m2. This study was reviewed and approved by the local regional Ethics Committee. The study adhered to the CONSORT guidelines in reporting this trial's results

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Clean wounds
* Informed consent
* Patients affected by Incisional and Ventral Hernia
* Elective surgery
* Hernia size between 3 e 7 cm
* BMI > 30 kg/m2

Exclusion Criteria:

* age < 18 years;
* Life expectancy < 24 months (as estimated by the operating surgeon), -
* Pregnancy
* Immunosuppressant therapy within 2 weeks before surgery
* Clean-contaminated and contaminated, dirty wounds
* Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2023 a series of 120 patients affected by Incisional Hernia with size between 3 to 10 cm, undergoing Intraperitoneal Onlay Mesh positioning in patients with BMI >30 kg/m2 in the clean wounds. The maximum enrollment time is 12 months.
  Clinical data will be collected in a prospective maintained electronic database, including patients' age, sex, body mass index (BMI), chronic corticosteroid use, albumin serum level, previous abdominal surgery or hernia, smoking habits, presence of diabetes mellitus (DM), presence of Chronic obstructive pulmonary disease (COPD). All the surgeries will be performed by experienced surgeons with at least 10 years of activity in the general surgery and emergency department with over 120 procedures of laparoscopically incisional hernia repair with insertion of non-absorbable and absorbable meshes. All patients enrolled in the study will be followed up by outpatient clinic controls performed by surgeons/surgical residents.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 1 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 3 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 6 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 12 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 24 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 36 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 1 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 3 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 6 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 12 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 24 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 36 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.

SECONDARY OUTCOMES:
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria
Number of patients affected by organ space infections | Within 30 days postoperatively
  Organ space infections according to Clavien-Dindo criteria
Number of patients affected by Surgical Site Occurence | Within 30 days postoperatively
  Surgical Site Occurence Reported according to the Ventral Hernia Working Group (VHWG) definitions
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 1 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale at 12 months.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale at 24 months.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pizza, MD, PhD, Principal Investigator — Azienda Sanitaria Locale Napoli 2 Nord
Locations (1):
- Francdesco Pizza, Napoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
All Individual Participant Data that underlie results in a publication